CLINICAL TRIAL: NCT05527626
Title: Chronic Kidney Disease - REAL Life Study in Alsace
Acronym: CKD-REAL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8517
Record Dates: First submitted 2022-08-30; First posted 2022-09-02 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Chronic Kidney Diseases
Keywords: Kidney; Chronic Disease; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Chronic Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic kidney disease (CKD) is a public health problem and affects about 10% of the world's adult population with a constantly increasing incidence. The approach to CKD in France is centered on access to replacement therapy (dialysis, renal transplantation), the cost of which amounts to 4 billion euros (data from the REIN registry).

Real-life data are essential to specify the characteristics of patients with chronic kidney disease and the factors associated with the evolution of CKD and the occurrence of complications in order to improve the management of CKD before the suppletion stage.

Since October 2019, CKD at the severe stage (stage 4) and at the non-dialysis end stage (stage 5) is subject to an annual flat fee (Article L. 162-22-6-2 of the Social Security Code). The reimbursement of these lump sums by the health insurance is subject to the collection and transmission of certain medical data by the establishments.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years)
* Subject included in the MRC package (GFR <30 ml/min/1.73 m2)
* Subject who has not expressed opposition, after information, to the reuse of his or her data for the purpose of this research

Exclusion criteria:

- Subject having expressed his opposition to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years) with a chronic renal disease
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Retroanalysis of the risk factors in patients with severe chronic kidney disease | Files analysed retrospectively from October 01, 2019 to February 31, 2027 will be examined
  Analysis of risk factors in patients with severe chronic kidney disease by retrospectively analyzing health data contained in patient medical records

CONTACTS AND LOCATIONS:
Overall Officials: Peggy PERRIN, MD, Principal Investigator — Service Néphrologie-Dialyse-Transplantation - CHU de Strasbourg - France
Locations (1):
- Service Néphrologie-Dialyse-Transplantation - CHU de Strasbourg - France, Strasbourg, France